CLINICAL TRIAL: NCT02156609
Title: HeartMate PHP™ CE Mark Clinical Investigation Plan
Acronym: HM PHP CE Mark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHPCEMark
Record Dates: First submitted 2014-05-29; First posted 2014-06-05 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: High Risk Percutaneous Coronary Intervention
Keywords: HeartMate PHP; HeartMate PHP CE Mark; Percutaneous coronary intervention; PCI; Percutaneous ventricular assist; Thoratec Corporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Percutaneous coronary intervention (Experimental): Percutaneous ventricular support with the HeartMate PHP during high risk percutaneous coronary intervention
  Interventions: Device: Percutaneous ventricular support with the HeartMate PHP

INTERVENTIONS:
Device: Percutaneous ventricular support with the HeartMate PHP — The HeartMate PHP device will be inserted percutaneously prior to the start of high risk coronary interventions (complex disease, reduced ejection fraction, etc.) to provide hemodynamic support,

SUMMARY:
The HeartMate PHP is a catheter-based pump designed to provide partial left heart circulatory support. The study will assess the safety and performance of the HeartMate PHP in supporting patients who are hemodynamically unstable, or at risk of being hemodynamically unstable, while undergoing percutaneous coronary interventions (PCI), such as coronary stent placement.

DETAILED DESCRIPTION:
The HeartMate PHP (percutaneous heart pump) is a catheter-based axial flow pump designed to provide partial left ventricular circulatory support. The primary objective of this prospective, nonrandomized, multi-center, open-label trial is to assess the safety and performance of the HeartMate PHP in supporting patients who are hemodynamically unstable, or at risk of being hemodynamically unstable, while undergoing percutaneous coronary interventions (PCI).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Patient presents with a non-emergent need for complex PCI with:

  1. an ejection fraction of ≤35% requiring hemodynamic support during the procedure, AND
  2. the heart team has determined that the patient is not an optimal surgical candidate, OR the patient elects not to undergo surgery
* Written, signed, and dated informed consent

Exclusion Criteria:

* Emergent PCI
* ST elevation myocardial infarction within 7 days of procedure
* Cardiac arrest within 7 days of procedure requiring CPR or defibrillation
* Hemodynamic support with the HeartMate PHP post-PCI is anticipated
* Cardiogenic shock (SBP <90 mmHg for >1 hour with either cool clammy skin OR oliguria OR altered sensorium OR cardiac index <2.2 L/min/m2)
* Mural thrombus in the left ventricle
* History of aortic valve replacement
* Documented presence of aortic stenosis (orifice area of 1.5cm2 or less)
* Moderate to severe aortic insufficiency (echocardiographic assessment of aortic insufficiency graded as 2 or higher)
* Severe peripheral vascular disease
* Abnormalities of the aorta that would preclude surgery, including aneurysms and significant tortuosity or calcifications
* Planned use of rotablator or atherectomy during the procedure
* Serum creatinine > 3.5mg/dL within 7 days of procedure
* Liver dysfunction with elevation of liver enzymes and bilirubin levels to ≥ 3x ULN or INR (Internationalized Normalized Ratio) ≥2
* Uncorrectable abnormal coagulation parameters
* Active systemic infection requiring treatment with antibiotics
* Clinically relevant stroke or TIA within 3 months of procedure. Patients with suspected stroke or TIA within 3 months of procedure must have documented absence of neurological infarction
* Uncontrollable allergy or intolerance to heparin, aspirin, clopidogrel, ionic and nonionic contrast media, or any other potentially required anticoagulants or antiplatelet therapy drugs
* History of heparin induced thrombocytopenia
* Patient is pregnant or planning to become pregnant during the study period
* Participation in another clinical study of an investigational drug or device that has not met its primary endpoint-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | Post procedure or at hospital discharge (whichever is longer), 30 days post procedure
  Primary Performance Endpoint:
  Freedom from hemodynamic compromise during PCI procedure defined as: Mean Arterial Pressure (MAP) not falling below 60mm Hg for more than 10 minutes during the PCI procedure and additional pressor medication is not required.
  Primary Endpoint will be evaluated at:
  * Post procedure or at hospital discharge (whichever is longer)
  * 30 days post procedure
Composite of Major Adverse Events (MAE) | Post procedure or at hospital discharge (whichever is longer), 30 days post procedure
  Primary Safety Endpoint:
  Composite of Major Adverse Events (MAE):
  * device-related cardiac death,
  * new Q wave myocardial infarction,
  * surgical intervention due to device complication or malfunction,
  * device-related access site complication requiring intervention or device-related limb ischemia,
  * cerebral vascular accident (CVA),
  * new or worsening aortic valve insufficiency,
  * major bleeding complication (BARC 3 or >),
  * severe hypotension
  Primary Endpoint will be evaluated at:
  * Post procedure or at hospital discharge (whichever is longer)
  * 30 days post procedure

SECONDARY OUTCOMES:
Secondary Endpoint | Post procedure or at hospital discharge (whichever is longer), 30 days post procedure
  Efficacy of hemodynamic support as measured by:
  * Maximal decrease in cardiac power output (CPO) from baseline
  * Changes in central venous pressure from baseline (CVP)
  * Changes in pulmonary artery pressure from baseline (PAP)
  * Changes in pulmonary capillary wedge pressure from baseline (PCWP)
  * Changes in cardiac output from baseline (CO)
  * Changes in cardiac index from baseline (CI)
Major Adverse Event Composites | Post procedure or at hospital discharge (whichever is longer), 30 days post procedure
  Individual components of the major adverse event composites

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Dudek, MD, Principal Investigator — Jagiellonian University
Locations (7):
- Instituto del Corazon, Bucaramanga, Colombia
- Erasmus Medical Center, Rotterdam, Netherlands
- Sanatorio Italiano, Asunción, Paraguay
- Poland (4):
  - Samodzielny Publiczny Szpital (The Prof. Leszka Gieca Upper-Silesian Medical Centre), Katowice
  - University Hospital in Krakow (John Paul II), Krakow
  - The Cardinal Stefan Wyszynski Institute of Cardiology, Warsaw
  - Slaskie Centrum Chorob Serca w Zabrzu (Silesian Center for Heart Disease), Zabrze